CLINICAL TRIAL: NCT01129037
Title: Goal Directed Fluid Management and Patient Outcome in Free Flap Reconstructive Surgery for Head and Neck Oncology: a Feasibility Randomized, Controlled Trial
Brief Title: Goal Directed Fluid Therapy in Free Flap Reconstructive Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UHN REB 09-0084BE
Record Dates: First submitted 2010-05-17; First posted 2010-05-24 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Head and Neck Cancer
Keywords: Oncology
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Goal directed fluid management (Other)
  Interventions: Other: Goal directed fluid management based on continuous monitoring of stroke volume

INTERVENTIONS:
Other: Goal directed fluid management based on continuous monitoring of stroke volume — Baseline SV measurement, repeated volume loading (VL) with aliquots of 250 ml HES until SV increased < 10% in response to receding VL: SV is optimized, no further VL required.

SUMMARY:
Wide excision of head and neck cancer with microsurgical free flap's reconstruction (FFR) results to a high cancer cure rate and a good functional recovery. However, this long complex procedure is accompanied with considerable complications. Excessive fluid administration during this type of surgery has been connected with poor results. There is growing evidence that goal-directed fluid management (GDFM) might improve the results in high-risk patients.

Hypothesis: Goal directed fluid management will reduce intraoperative fluid volume administered to patients undergoing head and neck reconstructive surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Signed informed consent

Exclusion Criteria:

* History CHF
* Severe valvular heart defects, intra cardiac shunts
* Irregular heart rhythm
* Allergy to hydroxyethyl starch solutions
* Coagulation abnormalities (INR>1.5, aPTT>40s, platelet count<100x10 9/L
* History of severe bleeding disorders
* Renal insufficiency with creatinine >200Umol/L
* Pregnant of nursing women
* History of skin disorders that are accompanied by chronic puritis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2010-07; Primary Completion 2012-05 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
The volume of fluid administered intraoperatively during reconstructive surgery for head and neck oncology | Initiation of surgery to end of surgery on average 8-10 hours

SECONDARY OUTCOMES:
Incidence of major complication and LOS | Post operative day 0 to hospital discharge
  Cardiovascular, respiratory, neurologic, thromboembolic, renal,liver, GI, sepsis,and surgical complications willl be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Leonid Minkovich, MD, Principal Investigator — Toronto General Hospital, UHN
Locations (1):
- Toronto General Hospital, UHN, Toronto, Ontario, Canada